CLINICAL TRIAL: NCT06564181
Title: The Relation Between Serum Zinc and Lupus Nephritis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Ashraf Anwar Abdelgalil, Principal investigator, Assiut University
Other Study IDs: Serum zinc and lupus nephritis
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to investigate the relation between serum zinc and lupus nephritis by search Prevalence of hypozincemia in lupus nephritis and Association between serum zinc and urea, serum creatinine, hemoglobin, estimated glomerular filtration rate (eGFR).

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic autoimmune disease affecting various organs including the skin, joints, kidneys, brain and heart...

Lupus nephritis (LN) is one of the most common severe organ manifestations of SLE . LN is clinically evident in 50-60% of patients with SLE , and it is histologically evident in most SLE patients, even those without clinical manifestations of kidney disease.

LN is associated with significant morbidity and mortality in SLE patients, as up to 20% of patients progress to end-stage renal disease (ESRD). The clinical manifestations of LN are variable, ranging from asymptomatic proteinuria to a myriad of manifestations associated with nephritic and nephrotic syndromes and ESRD.

Zinc is a vital micronutrient involved in numerous physiological processes including immune function, antioxidant defense, and cellular repair. It is a cofactor for over 300 enzymes and plays critical roles in DNA synthesis, protein production, and cell division. Zinc deficiency can impair immune function, increase oxidative stress, and hinder tissue repair, which are all relevant factors in autoimmune diseases like SLE, making its study in the context of LN particularly relevant.

However, further research is needed to fully understand the mechanisms and to develop evidence-based guidelines for zinc supplementation in lupus nephritis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lupus nephritis

Exclusion Criteria:

* other patients with other renal diseases .
* patients with other autoimmune diseases.
* patients on dialysis.
* patients with Diabetes mellitus.
* patients with liver diseases.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Patient with lupus nephritis .
  * patients with sex and age matching health control ( control group)
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hypozincemia in lupus nephritis Correlation between hypozincemia and urea , S. Creatinine and eGFR | 1/9/2024 - 1/9/2025
  Prevalence of hypozincemia in lupus nephritis

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Abdel Mawgoud, Dr, Study Director — Assiut University